CLINICAL TRIAL: NCT05751005
Title: The Impact of Collagen Peptide Supplementation on Joint Pain and Fat-Free Mass in Lifelong Athletes
Brief Title: Collagen Peptide Supplementation and Lifelong Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Tessenderlo Group (Unknown)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00000044
Record Dates: First submitted 2023-01-25; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Two different doses of collagen peptides versus placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This was a double blind study, in which investigators were not unblinded until all primary data end points were statistically analyzed. One person who was not involved in the study maintained the key until investigators were ready to be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen Supplementation 6 months (Experimental): Participants were randomized into one of three treatment groups for 6 months (Placebo, 10 g/d collagen peptides, or 20 g/d collagen peptides).
  Interventions: Dietary Supplement: Collagen Peptides vs. Placebo
- Collagen Supplementation 9 months (Experimental): Participants were randomized into one of three treatment groups (Placebo, 10 g/d collagen peptides, or 20 g/d collagen peptides) for additional 3 months after successful completion of the 6 month time point (total of 9 months).
  Interventions: Dietary Supplement: Collagen Peptides vs. Placebo

INTERVENTIONS:
Dietary Supplement: Collagen Peptides vs. Placebo — Participants were randomized into one of three treatment groups.

SUMMARY:
The aim of the current research is to evaluate the effects of 6 and 9 months of Solugel® supplementation on joint mobility, comfort, performance, body composition and related biomarkers of joint and bone health in older life-long athletes and physically active people. Doses of zero, 10, and 20 g per day for 6 or 9 months will be administered to determine, if any, is most effective at improving the previously mentioned outcomes.

DETAILED DESCRIPTION:
2.0 Objectives*

2.1 The aim of the current research is to evaluate the effects of 6 and 9 months of Solugel® supplementation on joint mobility, comfort, performance, body composition and related biomarkers of joint and bone health in older life-long athletes and physically active people. Doses of zero, 10, and 20g per day for 6 or 9 months will be administered to determine, if any, is most effective at improving the previously mentioned outcomes

2.2 We hypothesize that Solugel® at 10g and 20g will be more effective than the placebo supplement at all outcome measures. We also hypothesize that 20g will be more effective than 10g.

3.0 Background*

3.1 Very active individuals may describe joint discomfort as one negative aspect limiting their healthy lifestyles. Indeed, competitive swimmers (Wanivenhaus et al. Sports Health. 2012; 4:246-51) and those who partake in significant outdoor activity report substantial joint discomfort (Mranda et al. Osteoarthr Cartil. 2002; 10:623-30). This joint discomfort may be related to osteoarthritis (OA), a degenerative joint disease, presenting with focal and progressive loss of hyaline cartilage of joints with joint space narrowing. Current treatment for OA and joint pain include injectable corticosteroids and non-steroidal anti-inflammatory drugs. These modes of treatment are effective for reducing pain, however, they are not without serious long-term adverse effects including joint infection, nerve damage, possible tendon weakening, dyspepsia, ulcers, bleeding and other gastrointestinal complications.

In addition, very active individuals often complain of musculoskeletal injuries. Indeed, more than half of all sports injuries include sprains, ruptures, and damage to musculoskeletal tissue. The integrity of collagen-rich extracellular matrix that surrounds tendon, ligaments, and bone determines both the structure and function of these musculoskeletal tissues.

Nutritional interventions that strengthen these musculoskeletal tissues likely have a direct effect on injury prevention and rehabilitation. Indeed, supplementation with 5g or 15g of gelatin in subjects that performed high-intensity intermittent exercise bouts demonstrated improved collagen synthesis. In young athletic subjects, supplementation with 5g bioactive collagen peptides for 12 weeks demonstrated significant improvements in activity-related pain intensity compared to a placebo. The timing of collagen peptide intake in relation to improvements in functional outcomes is still not determined. Only one study to date has examined the influence of post-exercise collagen peptides compared to a placebo. The outcomes of this singular study demonstrated exceptional body composition improvements in elderly sarcopenic men. The increase in fat-free mass (FFM) and decrease in fat mass (FM) for the treatment group (FFM: +4.2±2.3 kg; FM: -5.4±3.1 kg) was significantly greater than the placebo group (FFM: +2.9±1.8kg; FM: -3.5±2.2 kg)). These changes in only 12 weeks were so pronounced that it warranted a letter to the editor by renowned protein researchers questioning the likelihood of such changes. To date, there has been no follow-up study to replicate these findings with regard to body composition.

Aging clearly exacerbates joint pain and worsens body composition resulting in less strength, less power, and decrements in exercise performance: an investigation using collagen peptides in life-long athletes over age 50 years is clearly warranted. Therefore, we aim to evaluate the effects of 9-months of Solugel® supplementation on joint mobility, comfort, performance, body composition and related biomarkers of health in older athletes.

4.0 Study Endpoints*

4.1 To determine the extent to which Solugel® can improve joint health as measured by a modified-Knee Injury & Osteoarthritis Outcome Score (mKOOS), and/or global & modified-Western Ontario and McMaster Universities Arthritis Index (WOMAC) subscales (discomfort, stiffness & function). Secondary outcome measures will include visual analog scale (VAS) questionnaires for overall/whole-body joint pain and changes in knee range of motion as assessed using a goniometer. Tertiary outcomes will include measures of cartilage synthesis and degradation (plasma IGF-1, P1NP, CTX, TGF-beta, MMPs), inflammation (plasma CRP, TNF-α), and bone formation and resorption (serum b-ALP).

To identify the extent to which Solugel® can improve body composition as measured with BIA and dual-energy x-ray absorptiometry (DXA) (fat mass, fat-free mass). In addition, bone mineral density (BMD) will be assessed (whole body, lumbar spine (L1-4) and left and right hip).

5.0 Study Intervention/Investigational Agent

5.1 Participants will be randomly assigned to one of three treatment groups: 1) placebo (maltodextrin); 2) 5g Solugel® + half serving of placebo; or 3) 10g Solugel®. Supplements will be consumed 2 times per day for 9 months. Compliance will be assessed at various time points throughout the duration of the study. Measurements will be taken at baseline, 1 month, 3 months, 6 months, and 9 months.

6.0 Procedures Involved*

6.1 To avoid risk of infection and spread of COVID-19, all participants will be screened for symptoms per the current CDC guidelines. PPE will be worn by all research personnel and participants, and six feet distancing will always be maintained when possible. All non-essential in person visits will also be moved to an online format. The facilities and equipment will be disinfected prior to study visits, and participants will be given the form HRP-502ic to update them on FSUs policies regarding mitigating the infection and spread of COVID-19.

Testing measures will include: Medical history questionnaire and aerobic fitness level (baseline only), anthropometrics, physical activity questionnaire (once per month), DXA scan, BIA, three day food records, pain questionnaire (once per month), range of motion (once per month), and blood sampling.

Over the span of the study, participants will be randomly assigned to receive one of the following treatments to be consumed 2 times per day: (1) Isocaloric placebo control (maltodextrin, PLA); (2) 5g Solugel® + half serving of PLA (LOW); (3) 10g Solugel® (HIGH). The supplements will be provided in identical packages and consumed with water. One month of the supplement will be provided at each visit. Compliance will be ensured via phone and email contact. A self-reported side-effects form will be completed monthly.

Baseline (0 months) Participants will arrive to the laboratory and complete screening questions, medical history questionnaires, physical activity questionnaires, pain questionnaires, informed consent documents, anthropometrics, DXA scan for bone density as well as body composition, BIA for TBW, three-day food records, range of motion testing, and blood sampling (20 ml).

Month 1 Participants will arrive to the laboratory and perform anthropometrics, DXA scan for body composition only, BIA for TBW, physical activity questionnaires, pain questionnaires, 3-day food records, and range of motion testing.

Months 2, 4, 5, 7, 8 Participants will arrive to the laboratory and perform pain questionnaires, physical activity questionnaires, and range of motion testing.

Month 3 Participants will arrive to the laboratory and complete screening questions, medical history questionnaires, physical activity questionnaires, pain questionnaires, informed consent documents, anthropometrics, DXA scan body composition only, BIA for TBW, three-day food records, range of motion testing, and blood sampling (20 ml).

Months 6 & 9 Participants will arrive to the laboratory and complete screening questions, medical history questionnaires, physical activity questionnaires, pain questionnaires, informed consent documents, anthropometrics, DXA scan for bone density as well as body composition, BIA for TBW, three-day food records, range of motion testing, and blood sampling (20 ml).

All measures are performed by trained study staff to monitor subjects for safety and to minimize risks.

6.2 The risk of adverse events from consumption of the supplement beverage is extremely minimal. Body composition and bone mineral density will be evaluated by DXA. This involves low exposure to radiation (less than 5 mREMs per DXA scan). Therefore, subjects undergoing the DXA scan can have a slightly increased cancer risk. By comparison, an x-ray of the spine is 70 mREM, a mammogram is 45 mREM, and a round trip transcontinental plane flight is 6 mREM. The risk of adverse events from the aerobic fitness test are minimal, blood draw may cause infection, localized bruising and discomfort, but all measures will be conducted by qualified personnel who will be present during all experimental trials to ensure proper procedures are followed. The risk of injury during the tests will be minimized by careful review of my medical history form, and no other assessments carry a risk of harm to participants.

6.3 Information obtained during the course of the study will remain confidential to the extent required by law. Participant names will not appear on any of the results. No individual responses will be reported in publication, only group responses. Confidentiality will be maintained by the assignment of a code number for each subject in which all data recorded will be based. The only record containing both the participant's name and code number will be kept by the principal investigator, Dr. Michael Ormsbee, in a locked drawer in his laboratory. All records will be destroyed after a minimum of five years.

7.0 Study Timelines*

7.1 Individual participant study duration is 6 or 9 months. The duration anticipated to enroll all study subjects is two years, and the estimated date for the investigators to complete this study is July, 2022.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 40-65 year.
* Perform greater than 4 hours per week of planned physical activity for the last 15 years.
* Report having periodic but sustained joint and/or musculoskeletal pain.
* Live in or near Tallahassee, FL.

Exclusion Criteria:

* Currently consuming collagen supplements (a 4 week washout period from the excluding supplement may be performed for the participant to be included).
* Currently using prescription pain medications (and cannot discontinue use during enrollment).
* Cortisone shot within the past 30 days (30 day washout period required).
* Smoking.
* Diagnosis of arthritis in the joints of interest (knee, hip, or shoulder joint).
* Diagnosis of autoimmune disorder.
* Initiation of hormone replacement therapy within the past 12 months.
* Uncontrolled medicated hypertension.
* Diagnosed kidney dysfunction.
* Allergies to milk or animal products.
* Surgery within the past 12 months.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Joint Health | 9 months
  Knee Injury and Osteoarthritis Outcome Score (KOOS). Scores are from 0 to 100, with a score of 100 being the best score, and a score of 0 being the lowest.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Science and Medicine, Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No